CLINICAL TRIAL: NCT02343991
Title: A Study to Evaluate the Safety and Feasibility of Blood-Brain Barrier Disruption Using Transcranial MRI-Guided Focused Ultrasound With Intravenous Ultrasound Contrast Agents in the Treatment of Brain Tumours With Doxorubicin
Brief Title: Blood-Brain Barrier Disruption Using Transcranial MRI-Guided Focused Ultrasound
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBB001; 215600 (Other: Health Canada)
Record Dates: First submitted 2015-01-12; First posted 2015-01-22 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transcranial ExAblate (Experimental): MR Guided Focused Ultrasound
  Interventions: Device: Transcranial ExABlate

INTERVENTIONS:
Device: Transcranial ExABlate — MR Guided Focused Ultrasound
  Other Names: ExAblate; TcMRgFUS

SUMMARY:
The purpose of this study is to evaluate the safety of BBB disruption using transcranial MRI-guided focused ultrasound in conjunction with an intravenous ultrasound contrast agent to increase the accumulation of doxorubicin in brain tumours and the adjacent brain using the ExAblate Transcranial system (220 kHz). Data will be collected to establish the basic safety of this type of treatment as the basis for later studies to evaluate its clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Men or women.
* Age between 18 and 70 years, inclusive.
* Able and willing to give informed consent.
* Size of the targeted portion of the tumour (i.e. prescribed ROT) is less than 2.5 cm in diameter (16 cm3). The non-targeted tumour tissue may exceed the targeted volume.
* Karnofsky rating 70-100
* ASA score 1-3.
* Able to communicate sensations during the ExAblate MRgFUS procedure.
* Able to attend all study visits (i.e., life expectancy of at least 3 months).
* At least 14 days passed since last brain surgery.

Exclusion Criteria:

* The sonication pathway to the tumour involves:

  i. More than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp ii. Clips or other metallic implanted objects in the skull or the brain, except shunts
* The subject presents with symptoms and signs of increased intracranial pressure (e.g., headache, nausea, vomiting, lethargy, and papilledema)
* Cardiac disease or unstable hemodynamics including:

  i. Documented myocardial infarction within six months of enrolment ii. Unstable angina on medication iii. Congestive heart failure iv. Left ventricular ejection fraction below the lower limit of normal v. History of a hemodynamically unstable cardiac arrythmia vi. Cardiac pacemaker
* Severe hypertension (diastolic BP > 100 on medication)
* Anti-coagulant therapy, or medications known to increase risk of hemorrhage, (e.g.:ASA, non-steroidal anti-inflammatory drugs (NSAIDs), statins)
* History of a bleeding disorder, coagulopathy or with a history of spontaneous tumour hemorrhage
* Abnormal level of platelets (< 100000), PT (>14) or PTT (>36), and INR > 1.3
* Documented cerebral infarction within the past 12 months
* TIA in the last 1 month
* Cerebral or systemic vasculopathy
* Insulin-dependent diabetes mellitus
* Immunosuppression (corticosteroids to prevent/treat brain edema are permitted)
* Known sensitivity to gadolinium-DTPA
* Contraindications to MRI such as non-MRI-compatible implanted devices
* Large subjects not fitting comfortably into the MRI scanner (generally >250 lbs)
* Difficulty lying supine and still for up to 4 hours in the MRI unit or claustrophobia
* Untreated, uncontrolled sleep apnea
* Positive pregnancy test (for pre-menopausal women)
* Known life-threatening systemic disease
* Severely impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2 and/or on dialysis
* Right to left or bi-directional cardiac shunt
* Previous full course of doxorubicin chemotherapy
* Allergy to eggs or egg products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-10; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Device and Procedure related adverse events | At the time of ExAblate transcranial procedure
  To evaluate the incidence and severity of adverse events (AEs) associated with the ExAblate transcranial treatment

SECONDARY OUTCOMES:
Severity of Device and Procedure related adverse events | At the time of ExAblate transcranial procedure
  To evaluate the incidence and severity of adverse events (AEs) associated with the ExAblate transcranial treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Mainprize T, Lipsman N, Huang Y, Meng Y, Bethune A, Ironside S, Heyn C, Alkins R, Trudeau M, Sahgal A, Perry J, Hynynen K. Blood-Brain Barrier Opening in Primary Brain Tumors with Non-invasive MR-Guided Focused Ultrasound: A Clinical Safety and Feasibility Study. Sci Rep. 2019 Jan 23;9(1):321. doi: 10.1038/s41598-018-36340-0. PMID 30674905